CLINICAL TRIAL: NCT05238545
Title: The Effect of Gluten-free Diet on Clinical Symptoms, Immune Parameters and Metabolome in Neurodegenerative Diseases With Alfa-synucleinopathy
Brief Title: The Effect of Gluten-free Diet on Parkinsonism
Acronym: GFREEPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General University Hospital, Prague (Other)
Collaborators: Czech Academy of Sciences (Other)
Responsible Party: Principal Investigator, Hana Brozova, Head of the movement disorder section in GUH Prague, General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NU21-04-00443
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease; Multiple System Atrophy; Non-celiac Gluten Sensitivity
Keywords: Parkinson Disease; Multiple system atrophy; Gluten-free Diet
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy | interventions — Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: Study groups in PD and MSA group with gluten-free diet and on regular gluten-containing diet. Randomization: patients will be randomized by diagnosis, age and disease duration, a numbered envelope in 1:1 ration to gluten-free diet group and regular gluten-containing diet group will be used.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PD gluten-free diet group (Experimental): Subjects with PD on gluten-free diet, ie. excluding all gluten-containing food during the day.
  Interventions: Other: gluten-free diet
- PD gluten-containing diet group (No Intervention): Subjects with PD on regular, gluten-containing diet, i.e. no restrictions during eating.
- MSA gluten-free diet group (Experimental): Subjects with PD on gluten-free diet, ie. excluding all gluten-containing food during the day.
  Interventions: Other: gluten-free diet
- MSA gluten-containing diet group (No Intervention): Subjects with MSA on regular gluten-containing diet, i.e. no restrictions during eating.

INTERVENTIONS:
Other: gluten-free diet — Diet excluding foods containing gluten.
  Arms: MSA gluten-free diet group; PD gluten-free diet group

SUMMARY:
Recent data suggest that the brain-gut axis, chronic intestinal inflammation and microbiome may contribute to the pathogenesis of neurodegenerative diseases with alfa-synucleinopathy, which include Parkinson's disease (PD) and Multiple system atrophy (MSA). Environmental factors e.g. diets, microbiome, metabolites and immune mechanisms may play important role in pathogenesis of these diseases. In the human arm of this project, the investigators will address effects of an anti-inflammatory gluten-free diet (GFD) on motor and non-motor symptoms as well as its effects on immune and metabolomic characteristics in patients with PD and MSA. In the mouse arm, the investigations will focus on the effects of GFD in chronic MPTP-induced mouse model of PD in various settings (e.g. in young or aged animals, with respect to the lengths of exposure to GFD). The chronic MPTP model will be used to assess the effects of GFD on adaptive and immune characteristics, and metabolic signatures. Using germ-free animals, the microbiome-dependency of the GFD-mediated effects may be determined. The anti-inflammatory gluten-free diet and its related mechanisms represent novel, promising and relatively straightforward approach in a search to improve symptoms of PD as well as MSA or even in their prevention.

DETAILED DESCRIPTION:
This project is based on two research lines, testing the effect of gluten-free diet in a patients with PD and MSA (a human prospective trial) and in the chronic MPTP (1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine)-induced mouse model of PD.

Research line 1. Assessments of effects of gluten-free diet (GFD) on clinical symptoms of Parkinson's disease (PD) and multiple system atrophy (MSA) in a prospective, controlled, randomized, rater-blinded human study. The goal of the research line 1 is to assess the effects of 12 months of administration of GFD on clinical symptoms of PD and MSA.

Research line 2. Effects of GFD on the development of PD in the chronic MPTP-induced mouse model of PD. The goal of the research line 2 is to study the effects of GFD in the chronic MPTP-induced mouse model of PD in order to evaluate its impact on clinical development of PD's features as well as immune and metabolomic characteristics that should shed more light on the possible mechanisms and potential novel treatment opportunities.

ELIGIBILITY:
Inclusion Criteria:

* subjects with establish diagnosis of PD in clinical stage 2-4 of Hoehn&Yahr scale or with establish diagnosis of MSA
* stable treatment for >4 weeks
* willing and able to give informed consent for participation in the study
* male and female subjects, aged 40 years or older
* able to understand and willing to comply with study procedures
* willing to avoid any other diet restrictions
* BMI 18-30

Exclusion Criteria:

* concomitant neurological, gastrointestinal or immunological disease
* diet restriction
* dementia affecting compliance
* acute psychiatric symptoms

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in severity of the clinical symptoms | Baseline, 1.5, 3, 6, 9, 12 and 13 months
  Scored by the MDS-Unified Parkinson's Disease Rating Scale (scores ranging from 0 to 260, higher scores indicate greater impairment) or Unified Multiple System Atrophy Rating Scale (scores ranging from 0 to 104, higher scores indicate greater impairment).

SECONDARY OUTCOMES:
Cognition change | Baseline, 1.5, 3, 6, 9, 12 and 13 months
  Scored by Montreal Cognitive Assessment (scores ranging from 0 to 30, lower scores indicate greater impairment).
Change in severity of the autonomic symptoms (Autonomic Scale for Outcomes in Parkinson's Disease) | Baseline, 1.5, 3, 6, 9, 12 and 13 months
  Scored by Autonomic Scale for Outcomes in Parkinson's Disease (scores ranging from 0 to 69, higher scores indicate greater impairment).
Change in spatio temporal parameters of the gait | Baseline, 1.5, 3, 6, 9, 12 and 13 months
  Investigated by GaitRite system
Quality of sleep change | Baseline, 1.5, 3, 6, 9, 12 and 13 months
  Scored by Pittsburgh Sleep Quality Index
Mood change | Baseline, 1.5, 3, 6, 9, 12 and 13 months
  Scored by Beck depression inventory (scores ranging from 0 to 63, higher scores indicate greater impairment).
Change in quality of life | Baseline, 1.5, 3, 6, 9, 12 and 13 months
  Scored by Quality of life questionnaire (scores ranging from 0 to 100, higher scores indicate greater impairment).

CONTACTS AND LOCATIONS:
Locations (1):
- GUHPrague, Prague, Czechia